CLINICAL TRIAL: NCT04896203
Title: Hypercoagulability Study Using Haemostatic Techniques in Patients With Inflammatory Bowel Disease
Acronym: EDGAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, María Dolores Martín Arranz, PhD, Principal Investigator, Hospital Universitario La Paz
Other Study IDs: PI-4182
Record Dates: First submitted 2020-11-24; First posted 2021-05-21 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Inflammatory Bowel Diseases; Thrombosis; Blood Coagulation Disorder
Keywords: Blood Coagulation; Blood CoagulationTests; Thrombelastography
MeSH Terms: conditions — Inflammatory Bowel Diseases; Thrombosis; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Ulcerative Colitis or Crohn's Disease patients, in remission according to inclusion criteria
  Interventions: Procedure: rotational thromboelastometry
- Group 2: Ulcerative Colitis or Crohn's Disease patients, with activity defined by the inclusion criteria
  Interventions: Procedure: rotational thromboelastometry

INTERVENTIONS:
Procedure: rotational thromboelastometry — Viscoelastometric method useful to study the kinetics of clot formation and fibrinolysis, providing a global information of both the cellular component and the pro and anticoagulant proteins, as well as the interactions between both components.

SUMMARY:
Descriptive study, in which the haemostatic profile of ambulatory patients with IBD will be analyzed by means of ROTEM and other techniques, such as the thrombin generation test and the study of platelet function by flow cytometry.

DETAILED DESCRIPTION:
Descriptive study, in which the haemostatic profile of ambulatory patients with IBD will be analyzed by rotational thromboelastometry (ROTEM) and other techniques, such as thrombin generation test and platelet function study by flow cytometry. The results of these measurements will be subsequently compared between the different IBD patient groups, stratified by activity and other risk factors, as well as with healthy controls, in order to define in which of these situations a significant prothrombotic risk exists, and which part of the coagulation cascade conditions that risk. After this, we will describe the incidence and prevalence of thromboembolic events in the follow-up of these patient groups. Finally, an attempt will be made to determine, according to the results of the study if any of the situations outside the classic recommendations would be subsidiary to receive chemoprophylaxis for the thromboembolic events.

The aim of this study is to determine the possible state of hypercoagulability of ambulatory patients with Inflammatory Bowel Disease, stratified according to the characteristics of their disease, by using ROTEM as well as the thrombin generation test. Platelet function will also be evaluated by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients diagnosed with UC according to ECCO criteria, in ambulatory follow-up in the IBD unit, stratified in remission and mild or moderate ambulatory management activity, determined by clinical (Simple Clinical Colitis Activity Index: SCCAI), biological (fecal calprotectin: CF), and/or endoscopic (Mayo Index) criteria: Remission: defined as a SCCAI < 2 and/or CF < 150 and/or May 0 index Activity: defined as an SCCAI >2, and/or CF > 150, and/or May Index >= 1 and <3.
* Patients diagnosed with CD according to ECCO criteria, in ambulatory follow-up in the IBD unit, stratified according to remission and mild or moderate ambulatory management activity, determined by clinical criteria (Harvey-Bradshaw index: HBI), biological criteria (CF) and/or endoscopic criteria (Simple Endoscopic Score-CD: SES-CD):

Remission: HBI < 5, and/or CF < 150, and/or SES CD < 3. Activity: HBI >=6 and <16, and/or CF > 150, and/or SES-CD >=3 (>4 if isolated ileal affectation) and <=15.

Exclusion Criteria:

* Patients with a previous history of venous or arterial thromboembolism
* Patients with recent hospitalization or surgery in the last 3 months.
* Women who are pregnant, undergoing treatment with oral contraceptives or who have received oral contraceptives in the last 3 months.
* Patients undergoing anticoagulation and/or active antiaggregation treatment
* Patients with severe activity criteria
* Patients with other concomitant conditions that favor thrombosis events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being followed in the Inflammatory Bowel Disease unit of the Hospital Universitario La Paz.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Platelet Function | Baseline
  Platelet activation will be evaluated by flow cytometry through analysis of fibrinogen (Fg) receptor activation and by exposure of P-selectin and CD63 on the surface of the platelets, in the basal state and after activation with thrombin receptor agonists.
Protein expression on Platelets Surface | Baseline
  Calibrated Automated Thrombogram (CAT) will be used to measure thrombin generation. CAT is a fluorimetric method that quantifies the amount of thrombin generated in a plasma sample after activation of the coagulation

SECONDARY OUTCOMES:
Thromboembolic Events | Baseline
  Thromboembolic events are one of the leading causes of mortality in Inflammatory Bowel Disease, and can occur in any of its subtypes. The most frequent are deep vein thrombosis of lower limbs and pulmonary thromboembolism.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Rueda García, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrd, Spain